CLINICAL TRIAL: NCT03237260
Title: An Open Label Single-arm Phase 4 Study of Vedolizumab in Subjects With Newly Diagnosed Active Ulcerative Colitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patient accrual
Sponsor: University of Pennsylvania (Other)
Collaborators: Takeda (Industry); Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 825665
Record Dates: First submitted 2017-07-26; First posted 2017-08-02 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vedolizumab 300mg (Experimental): vedolizumab open label
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Initiation: 300 mg at week 0, 2 and 6. Maintenance: Every 8 weeks after the sixth week at a fixed dose of 300 mg
  Other Names: entyvio

SUMMARY:
The purpose of this research study is to determine whether starting the drug vedolizumab earlier than its FDA approved use can lead to better control of UC then using older drugs that we have historically used to treat UC. Vedolizumab is FDA-approved to be used after initial Corticosteroid treatments have failed or other UC treatments have failed. We will study if using vedolizumab as an early treatment for your UC will allow you to get off corticosteroids and prevent UC from worsening and requiring surgery.

Vedolizumab is given intravenously initially every 2 weeks and then every 8 weeks.

DETAILED DESCRIPTION:
Based upon our published data, 53% of patients who require CS at the time of diagnosis of UC will be in CS free remission in the absence of colectomy by the end of 52 weeks. Early corticosteroids requirement after the diagnosis of ulcerative colitis diagnosis can predict a more severe long-term course of the disease. This work formed the basis of this research project. We had postulated that patients requiring steroids early in the course of their disease had worse prognosis than those who did not and should be treated more aggressively early in the course of their disease to prevent future complications like colectomy.

The current standard of care for treatment of UC in the VA is as follows:

At the time of diagnosis all the patients are started on a 5-ASA compound. Those patients who have very severe disease are concomitantly started on steroids. If they are very sick they are concomitantly started on an anti-TNF compound also with the goal of tapering them off steroids. Based upon response to therapy medications are adjusted. If there is no relief with 5-ASA compounds they can be started on steroids. For those on steroids and who cannot be weaned off steroids or are requiring multiple courses of steroids, they will have their therapy advanced to an anti-TNF or vedoluzimab. For those failing an anti-TNF they can be shifted to vedoluzimab. Thus, at the VA, vedoluzimab is available at the VA thru the non-formulary process. It is restricted to GI as 3rd line agent for UC. That is, it is used after oral agents fail and after anti-TNF agents (Humira® or Remicade®). The indications for Vedoluzimab use in the VA are as follows with regard to failure:

The patient has had adequate therapeutic trials of ONE of the following treatments, unless the patient has a contraindication, risk factor for serious adverse event*, or intolerance to the agent(s):

Criterion 1 is an option with or without therapeutic drug monitoring.)

A TNFI and an antimetabolite immunomodulator, separately or in combination. OR An initial and second TNFI, if therapeutic drug monitoring after secondary nonresponse to TNFI therapy indicates high titers of anti-TNFI antibodies.

OR

A TNFI, when either of the following apply:

Induction therapy with an agent from a different biologic class is needed to treat an inadequate response (with confirmed active inflammation / persistent disease) following TNFI induction therapy (i.e., primary nonresponse) and therapeutic drug monitoring shows therapeutic or high trough TNFI serum concentrations.

The patient lost response (i.e., secondary nonresponse not due to adverse reaction) to the initial TNFI in association with therapeutic or high trough TNFI serum concentration.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed active ulcerative colitis, defined as a Mayo Clinic score of 6 to 12
* Prior Sigmoidoscopy sub score of at least 2, and disease that extended 15 cm or more from the anal verge
* Must have required CS for treatment of their symptoms within 2 weeks of diagnosis and have not reached symptom adequate response and they still have moderate to severe disease, indicated by a Mayo score 6 - 12
* In subjects that enroll and are eligible to continue in the study, study drug needs to be started within 3 months of the subject starting corticosteroids

Exclusion Criteria:

* Currently treated with either anti-TNF therapy, immunomodulators or methotrexate due to the severity of their condition, making them not appropriate for vedolizumab
* Toxic megacolon, abdominal abscess, symptomatic colonic stricture, an increased risk of infectious complications
* An anticipated requirement for major surgery, colonic dysplasia or adenomas and malignant neoplasms
* Neurological disorders
* Pregnant or lactating females
* Clinical response to steroids prior to starting study drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
corticosteroid free remission as well as the absence of a colectomy | 52 weeks
  corticosteroid free remission as well as the absence of a colectomy

CONTACTS AND LOCATIONS:
Overall Officials: Nabeel Khan, MD, Principal Investigator — Assistant Professor of Clinical Medicine
Locations (2):
- United States (2):
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No